CLINICAL TRIAL: NCT02776397
Title: Relationship of Haptoglobin Phenotype to Vascular Function and Response to Vitamin E Supplementation in Patients With Diabetes Mellitus Type 2: The EVAS Trial
Acronym: EVAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tan Tock Seng Hospital (Other)
Collaborators: Lee Kong Chian School of Medicine, Nanyang Technological University (Unknown); National Medical Research Council (NMRC), Singapore (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: EVAS001 Version 4
Record Dates: First submitted 2016-05-12; First posted 2016-05-18 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-05

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Vitamin E; alpha-Tocopherol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Hp 2-2 Vitamin E (Active Comparator): The Haptoglobin 2-2 group randomised to Vitamin E
  Interventions: Dietary Supplement: Vitamin E
- Hp 2-2 Placebo (Placebo Comparator): The Haptoglobin 2-2 group randomised to placebo
  Interventions: Other: Placebo
- Non Hp 2-2 Vitamin E (Active Comparator): The Non Haptoglobin 2-2 group randomised to Vitamin E
  Interventions: Dietary Supplement: Vitamin E
- Non Hp 2-2 Placebo (Placebo Comparator): The Non Haptoglobin 2-2 group randomised to placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin E — Two hundred patients will be recruited to a pilot randomized controlled trial (RCT), stratified by Hp 2-2 phenotype status (100 Hp 2-2 and 100 non-Hp 2-2), and randomly allocated in a 1:1 ratio to either vitamin E 400 IU supplementation daily for 6 months or a placebo group. The trial will determine whether vitamin E improves the aforementioned surrogate markers in the Hp phenotype strata.
  Other Names: alpha tocopherol
  Arms: Hp 2-2 Vitamin E; Non Hp 2-2 Vitamin E
Other: Placebo — Placebo arm
  Arms: Hp 2-2 Placebo; Non Hp 2-2 Placebo

SUMMARY:
Relationship of haptoglobin phenotype to vascular function and response to Vitamin E supplementation in Patients with Diabetes Mellitus Type 2: The EVAS Trial

Specific Aims:

The phenotype haptoglobin 2-2 (Hp 2-2) is associated with higher oxidative stress, inflammation, LDL peroxidation and higher cardiovascular risk in patients with diabetes. We aim to determine whether Hp 2-2 phenotype is associated with surrogate markers of cardiovascular risk, inflammation, lipids and lipoprotein profile, oxidative stress, and endothelial cell (EC) apoptosis (in vitro study) in patients with diabetes in our population and whether vitamin E supplementation mitigates this risk.

Methods:

Screening Phase:

We will recruit 300 patients with diabetes mellitus type 2 (100 Chinese, 100 Malays and 100 Indians) and assess their Hp phenotype, surrogate markers of cardiovascular risk, inflammation, vascular biomarkers and lipids phenotype.

In vitro Study:

Plasma from 20 patients with Hp 2-2 phenotype and 20 patients with non Hp 2-2 phenotype will be studied in vitro using a haemodynamic lab-on-chip system to determine whether there is a difference in EC apoptosis between the two groups.

Randomisation Phase 200 patients will be recruited to a pilot randomized controlled trial (RCT), stratified by Hp 2-2 phenotype status (100 Hp 2-2 and 100 non-Hp 2-2), and randomly allocated in a 1:1 ratio to either vitamin E 400 IU supplementation daily for 6 months or a placebo group. The trial will determine whether vitamin E improves the aforementioned surrogate markers in the Hp phenotype strata.

Importance of proposed research to science and medicine:

This study allows us to understand the possible mechanism of cardiovascular risk in patients with Hp 2-2 phenotype and to see whether vitamin E supplementation reduces this risk in a pharmacogenomic targeted manner.

DETAILED DESCRIPTION:
1.0 Background and Clinical Significance 1.1 Introduction The incidence of Diabetes Mellitus type 2 (DM2) is growing rapidly globally and in Singapore. The main cause of increased morbidity and mortality in patients with DM2 is the development of microvascular and macrovascular complications. Although strict glycaemic control has been proven to reduce microvascular complications, the evidence is still lacking with regards to macrovascular complications. Accelerated atherosclerosis is the leading cause of increased mortality and morbidity in these patients. It is of paramount importance to assess novel targets to control atherosclerosis in patients with DM2 on top of conventional treatment. There is an unmet need to find new targets or markers predicting increased risk in patients with diabetes mellitus and we need to consider alternative treatments on top of conventional targets to reduce risk in these high risk group patients.

Patients with DM2 are not only at an increased risk for atherosclerosis, they also carry a greater extent of the disease burden. Endothelial dysfunction is considered the hallmark of the pathological insult inflicted on the blood vessels. Hyperglycaemia affects mitochondrial, enzymatic, and non-enzymatic pathways associated with the generation of reactive oxygen species (ROS), leading to decreased nitric oxide bioavailability and endothelial dysfunction, commonly demonstrated by reduced endothelium dependent vasodilatation and increased plasma levels of endothelium derived regulatory proteins. Moreover, DM2 patients have compromised antioxidant defenses in the form of low levels of the antioxidant enzymes and alpha-tocopherol (vitamin E), which may impede an adequate compensation for the increase in oxidative stress. Another role of oxidative stress in mediating the development of atherosclerosis has also been demonstrated in the oxidative hypothesis. In this model the most prominent target for oxidative modification is the LDL molecule. Oxidised LDL is not recognized by the LDL receptor but is readily taken up by the CD36 scavenger receptor pathway in macrophages leading to appreciable cholesteryl ester accumulation and foam cell formation. Oxidized LDL is proinflammatory, it causes inhibition of endothelial NO synthetase, promotes vasoconstriction and monocyte adhesion, and promotes platelet aggregation and thrombosis.

Hp Phenotype and Oxidative Tissue Damage

The haptoglobin (Hp) protein is an antioxidant due to its ability to neutralize the oxidative activity of haemoglobin (Hb). In humans, Hp is characterised by a genetic polymorphism with three structurally different phenotypes (Hp1-1, Hp 2-1 and Hp 2-2 which result from expression of two different alleles (Hp 1 and Hp 2) of the haptoglobin gene located on chromosome 16q22. The protein product of the Hp2 allele is an inferior antioxidant compared to Hp1 allele product. Hp 1-1 is a small molecule (86kDa) of well-defined structure, whereas Hp 2-1 is characterised by heteropolymers (86-300 kDA) and Hp 2-2 forms large macromolecular complexes (170-1,000 kDa).

The function of Hp is to bind free Hb released from red blood cells, which is released into the blood during the natural turnover of red blood cells. Free Hb is capable of causing considerable oxidative tissue damage as a result of its heme iron. However, whenever Hb is released into the circulation it immediately binds to Hp with extremely high affinity to form an Hp-Hb complex. This binding serves to inhibit the oxidative potential of Hb by preventing the release of heme iron from Hb. Hp is normally found in the blood in a more than 400-fold molar excess to free Hb and therefore Hp is capable of binding all of the Hb that is released during normal red blood cell turnover. Once Hb is bound to Hp it is rapidly cleared from the blood stream via the CD163 scavenger receptor expressed on monocyte/macrophages, however, formation and clearance of Hp-Hb complexes are impaired in Hp 2-2 phenotypes.

Iron derived from Hb can catalyse a number of oxidative reactions which can be inhibited by Hp .

1. Ferrous heme iron (Fe2+) can react with hydrogen peroxide to yield ferric Hb (Fe3+) and the highly reactive hydroxyl radical species. By abstracting a hydrogen atom from polyunsaturated fatty acids, hydroxyl radicals may initiate the process of lipid peroxidation.
2. Ferrous Hb (Fe2+) can also react with hydrogen peroxide to produce ferryl Hb (Fe4+), a highly unstable molecule which readily reacts with a second molecule of hydrogen peroxide to yield ferric Hb (Fe3+) and superoxide anion. The damaging effects of superoxide anion are two-fold: reduction of ferric iron (Fe3+) in Hb to ferrous iron (Fe2+), allowing for the production of additional hydroxyl radical as described in reaction 1, and dismutation of superoxide anion to produce hydrogen peroxide, again promoting the production of ROS.
3. Ferric Hb (containing Fe3+), also known as methaemoglobin, can spontaneously transfer its heme moiety resulting in heme entry into diverse lipophilic environments such as LDL or cell membranes. Once intercalated into its new lipid environment, heme iron can undergo reactions with hydrogen peroxide as described above or with adjacent lipid peroxides generating a free radical cascade and leading to extensive lipid oxidation.

   As a part of the Hp-Hb complex, Hp stabilizes heme in the heme pocket of Hb, and prevents Hb from causing oxidative injury . However, the degree to which Hp neutralizes the redox activity of heme iron differs among Hp types. This has been shown in a number of systems both in vitro and in vivo. For example, studies using linolenic acid showed that Hp 1-1 prevented oxidation (diene formation) as measured by an increase in absorbance at 232 nm to a greater extent than Hp 2-2 . Another study examined LDL oxidation due to heme transfer from Hb to LDL. Heme transfer was measured by quenching of the fluorescence signal emitted by dansylated LDL. It was found that Hp 1-1 was superior in preventing heme transfer from Hb as compared to Hp 2-2.

   Hp Phenotypes and Cardiovascular Risk Studies have shown that Hp 2-2 Hb complexes are also cleared less efficiently than non Hp 2-2 Hb complexes. In DM2 patients this phenomenon is more pronounced due to the downregulation of CD163, particularly in Hp 2-2 individuals. An impairment in anti-inflammatory macrophage signalling through a CD163/pAkt /IL-10 axis is also seen in Hp 2-2 patients.

   Hp-Hb deficient clearance in Hp 2-2 DM2 individuals results in increased Hp-Hb binding to Apo A1 on high-density lipoprotein (HDL-C), thereby tethering the pro-oxidative heme moiety to HDL. This renders it deficient in its ability to reverse transfer cholesterol from macrophages.

   The Hp 2-2 protein is less efficient at blocking heme transfer from Hb compared to Hp 1-1. Furthermore, the increase in heme transfer when Hb is glycosylated may provide a mechanistic explanation for the increase in cardiovascular disease seen in Hp 2-2 DM2.

   Hence Hp 2-2 phenotype is associated with decreased ability to bind with Hb, decreased clearance of Hp 2-2 Hb complexes, impairment in anti-inflammatory signalling pathway, increased LDL oxidation, renders HDL-Cholesterol inefficient and less efficient in blocking heme transfer from Hb to Hp 1-1 all leading to a higher cardiovascular risk. In diabetes patients where some of these pathways are also affected the synergetic effect of hyperglycaemia and haptoglobin phenotype is exacerbated leading to higher risk.

   In longitudinal studies done in other populations, it has been seen that Hp 2-2 genotype is associated with a 2-5 fold increased risk of incident CVD in individuals with DM. In particular the strong heart study the odds ratio of having CVD in DM with the Hp 2-2 phenotype was 2-5 times greater than in DM with Hp 2-1 phenotype (p=0.002). In the Munich Stent study a consecutive series of 935 treated diabetic individuals were followed up for one year after stenting for major adverse cardiac events. In this study the haptoglobin 2-2 phenotype was seen to be an independent predictor of major adverse cardiac events. In addition it has been seen that vitamin E provides substantial cardiovascular benefit to Hp 2-2 DM patients in one population (Israel-ICARE STUDY) and post-hoc analysis of the WHS (Women Health Study,) and HOPE study to see whether Vitamin E supplementation in subgroup of patients with the haptoglobin 2-2 phenotype influenced mortality showed a non-significant reduction in total mortality. This has not been widely adopted as larger trials, and on multiple populations, are needed to substantiate the association and benefits.

   Hp Phenotype and Ethnicity

   In a local study done in Singapore, it has been seen that the frequency of the Hp genes vary in the different ethnicities as follows :Chinese Hp1:0.330;Hp2:0.670;Hp0: 0.029; Malays:Hp1:0.298;Hp2:0.702 ;Hp0:0.004; Indians Hp1: 0.167;Hp2:0.833;Hp0:0.009. The distribution of the Hp frequencies has been seen to be at Hardy-Weinberg equilibrium in our population hence the expected prevalence of Hp 2-2 is around 30-40%. The Hp phenotypes will be determined by TaqMan analysis at the TTSH Research Laboratory.

   1.2 Haptoglobin genotypes and endothelial function

   Endothelial dysfunction has received increasing attention as a potential contributor to pathogenesis of vascular disease in DM. In DM2, the natural delicate balance in the release of contracting and relaxing factors by the endothelium is altered which contributes to further vascular and end-organ damage. Impaired endothelial function has been postulated to provide a final common pathway by which multiple risk factors exert their deleterious effects on cardiovascular health and has been established as a powerful surrogate marker for cardiovascular risk with one study showing even better predictability than the Framingham risk score . The EndoPAT 2000 device will be used as this has been established for estimation of endothelial function in a non-invasive manner.

   There are no direct studies done on looking at an association of Hp genotypes to endothelial function, in one pilot study wherein endothelial function was assessed using post-ischemic reactive hyperaemia and strain gauge plethysmography and expressed as maximal flow after an ischemic period, it was seen that Hp 2-2 patients with diabetes had worse endothelial function compared to non Hp 2-2 patients (450 +-50 versus 600+-40).

   1.3 Haptoglobin genotypes and CIMT (Carotid intima media thickness)

   In the Diabetes Heart study, genetic analyses of Hp genotypes showed an association between Hp 2-2 genotype and carotid intima media thickness (CIMT). These measurements will be made with the subject lying down, with the head extended and slightly turned opposite to the carotid examined, following the recommendations of the Mannheim CIMT consensus.Two investigators have estimated the CIMT in 23 individuals and a Bland-Altman plot was plotted and the limits of inter-user agreement was found to be within -0.1 to +0.1.

   1.4 Haptoglobin genotypes and aortic artery stiffness

   Although there are no direct studies done comparing Hp genotypes and aortic artery stiffness, one study was done wherein they evaluated the arterial elasticity of large and small arteries using pulse wave contour analysis method. The large artery elasticity index was lower in patients with Hp 2-2 compared with Hp 1-1 (8.4 +-2.3 ml/mmHg versus 12.6 +-4.1 ml/mmHg x 100; p<0.0001). In this study the small artery elasticity index was also significantly lower in patients with Hp 2-2 phenotype.

   Increased vascular stiffness has been seen early in the course of Diabetes Mellitus Type 2 using sphygmocor device. It is likely that this stiffness is related to endothelial dysfunction rather than structural vascular alterations-this in turn suggests that it is reversible. Aortic pulse wave velocity (PWV), a measure of aortic distensibility, has also been seen to predict mortality in patients with diabetes independently of known confounding factors. The SphygmoCor Xcel device to estimate the aortic artery stiffness using the carotid to femoral pulse wave velocity and central aortic pressure will be used. The investigators will estimate the pulse wave velocity in 20 individuals in order to establish the limits of agreement using the Bland-Altman plot before starting the study.

   1.5 Haptoglobin genotypes and vascular markers

   Vascular cell adhesion molecule-1 (VCAM-1) and intercellular adhesion molecule-1 (ICAM-1) are proteins expressed on the surface of activated endothelial cells (ECs) and expressed in early atherosclerosis. These markers have been evaluated and considered good markers of endothelial dysfunction because part of the protein is shed in the circulation and can be detected in peripheral plasma.

   1.6 Haptoglobin genotypes and phenotyping of plasma lipids

   Hp 2-2 phenotype has been associated with higher oxidised LDL concentrations, which is primarily involved in atherosclerosis. The concentrations of Apo-A1 HDL is also known to be higher in this group of patients. Hp 2-2 phenotype may also be associated with higher Lp(a) concentrations putting these patients at higher cardiovascular risk. Detailed phenotyping of plasma lipids using proteomics to look for novel associations will be done.

   1.7 Haptoglobin genotypes and Oxidative Stress

   It is known that Hp 2-2 genotype confers a higher oxidative stress on the endothelium. The total oxidative potential will be calculated as the Oxidative-INDEX. Two tests will be done as follows to calculate this index. This index has been established as a good estimate of the overall oxidative stress.
   1. d-ROMs test: This test will be performed on serum samples by using automated d-ROMs method. (Vassalle C, Pratali L, Boni C, Mercuri A, Ndreu R. An oxidative stress score as a combined measure of the pro-oxidant and anti-oxidant counterparts in patients with coronary artery disease. Clin Biochem 2008;41:1162-7)
   2. FRAP (ferric reducing ability of plasma - a measure of the ability of the plasma to prevent damage to vessels) and d-ROMs (derivatives for the Reactive Oxygen Metabolites) test will be used to calculate the oxidative stress score.

   Other markers of oxidative stress will also be measured such as glyoxal, methylglyoxal, asymmetric dimethylarginine and homoarginine.

   1.8 Haptoglobin genotypes and retinal Arteriovenous index

   The presence of retinal microvascular abnormalities especially arterial constriction and venular dilatation has been associated with an increased cardiovascular risk and has been associated with endothelial dysfunction and inflammation.Currently there are no studies looking at the relationship between Hp genotypes and retinal arteriovenous (AV) index. . Prior to the investigations, eye drops will be instilled to dilate pupils for fundus examination and to lubricate the cornea. Retinal imaging will be done for the subjects at the eye clinic. If patients do not wish to participate in the retinal imaging, they may choose to opt out from the retinal imaging test.

   2.0 Vitamin E, haptoglobin phenotype and cardiovascular risk reduction

   While functional differences between Hp1 and Hp2 allelic protein products particularly in DM can explain the differences in susceptibility to complications in the Hp 2-2 individuals from non Hp 2-2 individuals, the main reason of unique benefit from vitamin E is that redox active Hb is associated with HDL only in Hp 2-2 DM individuals. In patients with DM decreased Hp-Hb complexes results in increased Hp-Hb binding to Apo-A1 on high-density lipoprotein (HDL), thereby tethering the pro-oxidative heme moiety to HDL. HDL in Hp 2-2 DM individuals is deficient in its ability to stimulate the reverse transfer of cholesterol from macrophages. Besides these, the Hp phenotype 2-2 is associated with increased oxidative stress due to deficient clearance of free radicals and increased LDL peroxidation.

   Vitamin E is a potent antioxidant with anti-inflammatory properties. It significantly alleviates the condition of oxidative stress by both its potent free radical scavenging properties and by interacting directly and strongly with the antioxidant enzymes. Vitamin E supplementation in humans and animal models has shown to decrease lipid peroxidation, superoxide production and decreasing the expression of scavenger receptors (SR-A and CD36) which are particularly important in the formation of foam cells. Although vitamin E has not been proven to be useful in reducing cardiovascular risk in the general population, it has been useful in patients with Hp 2-2 phenotype with DM, both conditions which increase oxidative stress substantially in studies done in one population.

   There have been only three interventional randomized controlled trials (RCTs) in which the only antioxidant which the DM participants received was vitamin E and in which the Hp type of study participants was determined. The ICARE study was the only RCT aimed to evaluate vitamin E in DM patients for which Hp genotype was prospectively collected. In this study, 1,434 DM individuals > or = 55 years of age with the Hp 2-2 phenotype were randomised to vitamin E (400 IU/day/placebo). The primary composite outcome was significantly reduced in individuals receiving vitamin E (2.2%) compared to placebo (4.7%, p=0.001) at 18 months after initiation of the trial when it was terminated. Additionally, blood samples from a subset of patients recruited for the WHS and HOPE studies were analysed for Hp polymorphism, and the outcomes reassessed according to the patient's Hp type. In all these studies, a higher risk of cardiovascular events was seen in Hp 2-2 individuals and a benefit to vitamin E supplementation was seen in this group.

   2.1 Justification for dose and duration of vitamin E (alpha-tocopherol).

   We will be using vitamin E 400 IU per day and matched placebo. We will commission the company Beacons who will prepare the vitamin E capsules (400 IU) and the matching placebo capsules. Vitamin E preparation will be the natural tocopherol which occurs in the RRR-configuration. We will give vitamin E 400 IU for 6 months as most studies using surrogate markers of cardiovascular risk has seen an improvement in 6 months after supplementation. Moreover, in the ICARE study mentioned above an improvement in cardiovascular outcome was seen at 18 months thus suggesting that 6 months should be adequate duration to see an improvement in surrogate markers of cardiovascular risk.

   The eight forms of vitamin E are divided into two groups; four are tocopherols and four are tocotrienols. They are identified by prefixes alpha- (α-), beta- (β-), gamma- (γ-), and delta- (δ-). alpha-tocopherol is the most abundant form in nature, known to have the highest biological activity based on fetal resortion assays and reverses vitamin E deficiency symptoms in humans. Natural tocopherols occur in the RRR-configuration only. The synthetic form contains eight different stereoisomers and is called 'all-rac'-α-tocopherol.

   Vitamin E is found in its natural form in vegetable oils (wheat germ, sunflower, safflower, corn and soybean oils), nuts (almonds, peanuts and hazelnuts), seeds (sunflower seeds), green leafy vegetables (spinach and broccoli) and fortified breakfast cereals, fruit juices, margarine and spreads. The institute of Medicine recommended intakes for individuals is about 15mg/day. The highest safe level of vitamin E supplements for adults is 1,500 IU/day for natural forms of vitamin E, and 1,000 IU/day for the man-made (synthetic) form. Popular vitamin E supplements available includes, D-alpha tocopherol which is derived from natural oils. Commercially available vitamin E supplements usually contain only alpha-tocopherol provided either unesterified or as the ester of acetate, succinate or nicotinate. In humans, free and esterified alpha-tocopherol have the same bioavailability. Supplements can contain either the natural RRR-or synthetic (all-rac) alpha-tocopherol. The biological activity of natural RRR alpha-tocopherol is higher than that of synthetic all-rac-alpha-tocopherol and other natural forms of vitamin E.

   Both oxidative stress and individual genetic makeup contribute to vitamin E homeostasis in humans and this may be responsible for the variable clinical effects seen in improvement of clinical variables in clinical trials. Vitamin E is absorbed in the intestine, enters the circulation via the lymphatic system where absorbed together with lipids, it is packed into chylomicrons and transported to the liver. After passage through the liver, only alpha-tocopherol preferentially appears in the plasma and most of the other forms of vitamin E is preferentially metabolised and either secreted in the bile or not taken up and excreted in the faeces. In the liver, hepatic alpha-tocopherol transfer protein (α-TTP) specifically sorts out the α- form with the 2R-stereoisomers. Plasma RRR-α-tocopherol incorporation is a saturable process. Plasma levels of RRR-α-tocopherol cease to increase at approximately 80 μM despite increasing dosages of vitamin E supplementation of up to 1,320 mg all-rac-α-tocopherol per day. This is likely secondary to the rapid replacement of circulating with newly absorbed α-tocopherol and kinetic analyses demonstrates that the entire pool of α-tocopherol is replaced daily. In humans, the preferential accumulation of α-tocopherol in the body is dependent upon both a functional α-TTP and increased metabolism and excretion of non-α-tocopherols. The alpha-tocopherol transfer protein regulates whole-body distribution and concentrations of vitamin E by controlling the secretion of vitamin E from the liver. It has been seen that the expression of the alpha-tocopherol transfer protein gene can be induced by oxidative stress and hypoxia, by agonists of the nuclear receptor PPARα and RXR, and by increasing cAMP levels. This is mediated by an already present transcription factor called cAMP response element-binding (CREB) transcription factor. Single-nucleotide polymorphisms that are commonly found in healthy people drastically affect promoter activity.

   Various doses of vitamin E ranging from 400 IU to 2,000 IU have been used in clinical trials. The institute of medicine, USA suggests a recommended dietary intake (RDA) of 15-1,000 mg/day (1 mg =1.5 IU; 22.5-1,500 IU/day). We are using a dose of 400 IU for six months. There is no evidence of adverse effects if taken within the RDA, However there may be haemorrhagic toxicity in high doses especially in patients on anticoagulants. Hence we will be excluding patients on anticoagulants.

   3.0 Statistical Considerations

   3.1 Sample size calculation: The overall estimated sample size for the study is 300 patients. The required sample size of 100 for each Hp phenotype stratum of the RCT phase is based on: 5% type I error; 90% power; the assumption that vitamin E is expected to have at least a moderate effect, represented by a standardized effect size (mean difference/pooled-standard error) of 0.5, on each risk marker; two sample t-test with equal variance; and a 15% drop out rate. Assuming 35% prevalence of Hp 2-2 in our population, we need to screen 300 patients to recruit 100 Hp 2-2 phenotype patients.

   Assuming a mean difference on RHI of 0.25 units with corresponding standard deviation (SD) of 0.3 - yielding a standardized effect size of 0.25/0.3 = 0.83 as minimal difference in RHI seen in another study. We did not adjust for multiple testing/comparisons due to the pilot nature of the RCT, as well as the exploratory nature of the study in general.

   The sample size for the in vitro study is constrained by limited resources. Nevertheless, simulation results based on a two-sided Wilcoxon Signed-Ranked test, 5% type I error, a correlation between pairs of 0.5, and 5000 Monte Carlo simulation samples indicate that 20 pairs provide adequate power to detect moderate to large standardized effect sizes (M1).

   Randomisation will be done electronically through the web - a centralized password-protected intranet website to ensure that the patients are randomised the moment they are eligible for the trial (strictly sequential). A blocked randomisation schedule will be employed, in blocks of 10, for the study based on a 1:1 allocation ratio. The dedicated password-protected site will then allocate a unique patient trial number which will correspond to the treatment numbers labelled in the medication boxes. Following randomisation, the first dose will be administered to the patient.

   3.2 Data handling and statistical analyses: Data Handling All relevant will be collected using appropriate well-designed study data-collection forms at each visit and telephone follow up assessment. All study data will be stored in a study database assessable only to data entry and data validation study personnel.

   Statistical Analysis Plan Data on baseline demographic and clinical variables as well as risk markers will be summarized by Hp phenotypes and overall to provide insight on potential associations. Binary data will be summarized using frequency and proportions. Chi-square test and Fisher exact test will be used to evaluate relevant associations (including benefits of vitamin E), and if necessary logistic regression will be used to characterize associations while adjusting for potential confounders. Continuous variables will be summarized using means (standard deviations) or median (range) as deemed appropriate. Two sample t-test or Mann-Whitney test will be used to evaluate relevant associations and generalized linear models will be used to characterize associations while adjusting for potential confounders. Generalized linear models are considered as they can accommodate non-normal (asymmetric) data or log-normal data (such as laboratory data) if necessary. Separate tests and models will be performed for each relevant outcome.

   Data from the in vitro study will be summarized similarly as described in the preceding paragraph, by Hp 2-2 phenotype status and vitamin E concentrations. Wilcoxon Signed-Ranked test will be used to evaluate the benefits of vitamin E between Hp phenotype groups by concentrations. Mann-Whitney and Jonckheere-Terpstra test will be used to evaluate the concentration-benefit relationship of vitamin E by Hp phenotype groups. Generalized linear mixed models will be employed to explore various trends and associations while accounting for (i) the matching of Hp 2-2 and non Hp 2-2 patients, (ii) repeated assessment within a patient by vitamin E concentration, (iii) adjusting for potential confounders, and (iv) adjusting for potential non-normality (asymmetry) of the data by using other appropriate distributions such as log-normal or gamma distributions. An overall analysis of the data from in vitro study will be done.

   Bland-Altman analysis will be used to estimate and evaluate the limits of agreement for the agreement and reliability studies. Where appropriate, a mixed model approach will be used to estimate and evaluate the relevant reliability coefficients.

   5.0 Clinical Significance

   If an association is seen between Hp 2-2 phenotype with cardiovascular risk, this group of patients can be targeted for vitamin E treatment on top of statins and other conventional treatment to reduce the cardiovascular risk. Future large scale nation-wide RCT can be planned to see whether vitamin E treatment helps to reduce the risk in this group of patients. Conducting such studies in a multi-ethnic population is imperative as it provides insight on the consistency and generalizability of the expected benefits.

ELIGIBILITY:
Inclusion Criteria:

Study patients should meet the following criteria for inclusion in the study:

1. 100 Chinese, 100 Malays, 100 Indian patients with DM2
2. Age 21-80 years
3. Able to give informed consent
4. Stable diabetes, blood pressure and hyperlipidaemia medications (a 25% dose adjustment is allowed) in the last three months
5. For eligibility to be randomized: HbA1c should be 10% inclusive or below at time of randomisation
6. Blood Pressure should be less than 180/120 mm Hg at time of recruitment
7. Non-smokers or discontinued smoking at least 6 months ago
8. No h/o previous myocardial infarction, previous cerebrovascular accident inclusive of haemorrhage and infarction, or h/o of peripheral amputation or bypass procedures

Exclusion Criteria:

1. Inability to give informed consent
2. Pregnant subjects
3. Patients hospitalized for any condition less than 1 month from enrolment
4. Patients having any recent infections or symptoms suggestive of any systemic infection in the last 2 weeks
5. Myocardial Infarction or stroke within 6 months before enrolment
6. Patients with creatinine concentrations >200 µmol/L or eGFR<30 µmol/L
7. Patients on anticoagulants such as warfarin
8. Known allergy to vitamin E
9. Current smokers
10. h/o previous myocardial infarction, previous cerebrovascular accident inclusive of haemorrhage and infarction, or h/o of peripheral amputation or bypass procedures
11. Patients on immunosuppressive agents or corticosteroids for other conditions
12. Presence of concomitant malignancies or rheumatological conditions at the time of recruitment
13. Patients taking orlistat & cholestyramine

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2015-06; Primary Completion 2018-06 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Endothelial function | 6 months
  Measured as Reactive hyperemia index using RHI-EndoPAT
Aortic artery stiffness | 6 months
  Measured as pulse wave velocity using the sphygmocor device
Carotid Artery Intima Media Thickness | 6 months
  Measured as CIMT (average) in mm.
Inflammation | 6 months
  Measured as hs-CRP
Oxidative Stress | 6 months
  Measured as oxidative stress index

SECONDARY OUTCOMES:
Glycemic status | 6 months
  Measured as HbA1c
Retinal arteriovenous index | 6 months
  Measured as ratio between retinal arterial diameter and venous diameter as retinal AV index
Non HDL-Cholesterol | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Rinkoo Dalan, MBBS, FRCP(Edin), Principal Investigator — Senior Consultant
Locations (1):
- Tan Tock Seng Hospital, Singapore, Singapore, Singapore

REFERENCES:
- [Background] Levy AP, Hochberg I, Jablonski K, Resnick HE, Lee ET, Best L, Howard BV; Strong Heart Study. Haptoglobin phenotype is an independent risk factor for cardiovascular disease in individuals with diabetes: The Strong Heart Study. J Am Coll Cardiol. 2002 Dec 4;40(11):1984-90. doi: 10.1016/s0735-1097(02)02534-2. PMID 12475459
- [Background] Milman U, Blum S, Shapira C, Aronson D, Miller-Lotan R, Anbinder Y, Alshiek J, Bennett L, Kostenko M, Landau M, Keidar S, Levy Y, Khemlin A, Radan A, Levy AP. Vitamin E supplementation reduces cardiovascular events in a subgroup of middle-aged individuals with both type 2 diabetes mellitus and the haptoglobin 2-2 genotype: a prospective double-blinded clinical trial. Arterioscler Thromb Vasc Biol. 2008 Feb;28(2):341-7. doi: 10.1161/ATVBAHA.107.153965. Epub 2007 Nov 21. PMID 18032779
- [Background] Blum S, Vardi M, Levy NS, Miller-Lotan R, Levy AP. The effect of vitamin E supplementation on cardiovascular risk in diabetic individuals with different haptoglobin phenotypes. Atherosclerosis. 2010 Jul;211(1):25-7. doi: 10.1016/j.atherosclerosis.2010.02.018. Epub 2010 Feb 21. No abstract available. PMID 20223458
- [Background] Levy AP, Gerstein HC, Miller-Lotan R, Ratner R, McQueen M, Lonn E, Pogue J. The effect of vitamin E supplementation on cardiovascular risk in diabetic individuals with different haptoglobin phenotypes. Diabetes Care. 2004 Nov;27(11):2767. doi: 10.2337/diacare.27.11.2767. No abstract available. PMID 15505023
- [Background] Saha N, Ong YW. Distribution of haptoglobins in different dialect groups of Chinese, Malays and Indians in Singapore. Ann Acad Med Singap. 1984 Jul;13(3):498-501. PMID 6517517